CLINICAL TRIAL: NCT01483482
Title: Neither Operative Nor Non-operative Approach is Superior Treating Displaced Midshaft Clavicle Fractures: a Randomised Clinical Trial
Brief Title: Treatment of Displaced, Midshaft Clavicle Fractures. Sling or Plate?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ilija Ban, Principal Investigator, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORH-IB-0001
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Acute, Displaced Midshaft Clavicle Fractures
Keywords: clavicle fractures; midshaft clavicle fractures; conservative treatment; surgical treatment; functional outcome; clinical assessment; adults
MeSH Terms: interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative treatment (Other): The group allocated to conservative treatment is treated with a simple sling. The sling is removed when the patient is pain free.
  The first 6 weeks max 1 kg of weight-bearing is allowed and the patient is instructed to restrict movement of the arm to the level of the shoulder.
  Interventions: Procedure: Conservative Treatment
- Surgical treatment (Other): Patients allocated to surgical treatment are operated with a superior locking plate.
  The first 6 weeks max 1 kg of weight-bearing is allowed and the patient is instructed to restrict movement of the arm to the level of the shoulder.
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Conservative Treatment — Simple Sling
  Arms: Conservative treatment
Procedure: Surgical treatment — Superior Locking plate
  Arms: Surgical treatment

SUMMARY:
Clavicle fractures are frequent and represent somewhere between 5 and 10% of all fractures seen in orthopedics.

There is no consensus concerning the best treatment of acute, displaced, midshaft clavicle fractures. Conservative treatment has, traditionally, been the preferred treatment but recent studies have shown higher incidences of non-union and symptomatic malunion associated with conservative treatment. Primary surgery has in several studies been associated with high success rates and few complications but there is no compelling evidence towards superior results after primary surgery.

The objective of this randomized study is to compare conservative treatment (sling) with primary surgery (locking plate) of acute, displaced, midshaft clavicle fractures.

DETAILED DESCRIPTION:
Conservative treatment has been the preferred treatment for midshaft clavicle fractures, whether the fracture is displaced or undisplaced. The background for this comes from two large studies done in the 60s. C. Neer (2235 patients) and C. R Rowe (566 patients) showed respectively in 1960 and 1968 that patients with a clavicle fracture, even with larger fracture displacements, had few symptoms when the fracture is healed and that the incidence of non-union is below 1%. Both studies have been criticized for including children and adolescents where the healing potential is significantly larger than in adults and that their results are based purely on surgical and radiologic endpoints and no patient-reported outcome measurements were used.

Clavicle fractures are frequent and represent somewhere between 5 and 10% of all fractures seen in orthopedics. The incidence of clavicle fracture is somewhere between 29 and 64 per 100000 per year. Fracture of the clavicle most frequently occurs in young men and the male-to-female distribution is 2.6:1. Between 70 and 80% of all clavicle fractures are localized to the middle part of the clavicle and of these, most fractures are displaced. Midshaft clavicle fracture is defined as a fracture in the middle 3/5 parts of the clavicle (lateral boundary is a vertical line from the base of processus coracoideus and medial border is a vertical line from the middle of the first rib).

Recent studies have shown higher incidences of non-union, especially when the fracture is displaced and a shortening of two cm or more occurs. Malunion, that was previously not considered clinically important, appears in several resent studies to be associated with profound symptomatic shoulder problems. One study reported that up to 30% of the displaced clavicle fractures that healed with malunion results in profound symptoms and discomfort of the shoulder.

Surgery, with plate osteosynthesis of the displaced clavicle fracture, has in several studies been associated with a high success rate and few complications. To date only one randomized trial comparing conservative treatment with plate osteosynthesis of the displaced midshaft fracture has been done. This Canadian multi-center study from 2007, where 132 patients were randomized (111 patients completing), concludes that there is a small significant improvement in functional outcome in patients where the fracture has been osteosynthesised compared with conservative treatment. This study recommends surgery of displaced fractures in active patients.

Recently two review articles have questioned the results from the Canadian study because it is unclear whether the poorer functional outcome in the conservatively treated group is due to the non-unions in this group (14.2%). They both conclude that there is an estimated risk of overtreatment as a numbers-needed-to-treat analysis estimates the 9 operations is needed to prevent 1 non-union.

Though the evidence for surgical intervention over conservative treatment for displaced midshaft clavicle fractures still is controversial it seems that more and more patients are treated with primary operative intervention.

Because of this tendency there is a need to validate whether operative intervention with a clavicle plate is superior or not compared to the conservative treatment for displaced midshaft clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* The patient can not have any medical untreated illness : only ASA 1-2
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.
* The patient is expected to be able to follow the postoperative controls.

Exclusion Criteria:

* Multitrauma patient
* Other simultaneous fractures
* Former surgery of the shoulder or clavicular.
* Former chronic illness of the shoulder
* Pathological or open fractures
* Associated nerve or vessel damage of the affected arm.
* Fractures older than 3 weeks (21 days)
* Patients with drug(alcohol abuse where it is not expected that the patient i able to complete the follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 12 month follow-up
  Constant score and DASH score is used to evaluate the functional score at 6 weeks, 6 months and 12 months.

SECONDARY OUTCOMES:
Clinical assessment | 12 month follow-up
  Clinical and radiological assessment is done at 6 weeks, 6 months and 12 months of follow-up. Non-union, symptomatic manlunion,surgical complication (infection, hardware failure) is registered.

CONTACTS AND LOCATIONS:
Overall Officials: Ilija Ban, MD, Principal Investigator — University Hospital of Hvidovre; Anders Troelsen, MD, PhD, Study Director — University Hospital of Hvidovre
Locations (1):
- University Hospital of Hvidovre, Hvidovre, Denmark